CLINICAL TRIAL: NCT05173441
Title: A Randomized, Double-blind, Placebo-controlled Phase II Exploratory Clinical Trial to Evaluate the Efficacy and Safety of Human COVID-19 Immunoglobulin (pH4) for Intravenous Injection (COVID-HIG) in the Treatment of Patients With COVID-19
Brief Title: Human COVID-19 Immunoglobulin (COVID-HIG) Therapy for COVID-19 Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sinopharm Wuhan Plasma-derived Biotherapies Co., Ltd. (Industry)
Collaborators: China National Biotec Group Company Limited (Industry); Beijing Tiantan Biological Products Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Beijing Tiantan Biological Products Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: COVID-19-IVIG-201
Record Dates: First submitted 2021-11-23; First posted 2021-12-30 (Actual); Last update posted 2022-01-03 (Actual); Status verified 2021-12

CONDITIONS: COVID-19
Keywords: COVID-19; immunoglobulin; COVID-HIG; SARS-CoV-2; 2019nCov; hyperimmune globulin; Coronavirus disease 2019; passive immunotherapy; therapeutic
MeSH Terms: conditions — COVID-19 | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High Dose Group (Experimental): Standard of care (SOC)+high dose COVID-HIG. COVID-HIG will be administered via intravenous infusion. once a day, for three consecutive days (Day 0, day 1, and Day 2). And it could be administered again for 1-2 days according to the clinical improvement of subjects, and the total number of infusions should not exceed5 times.
  Interventions: Biological: Human COVID-19 immunoglobulin (pH4) for intravenous injection
- Low Dose Group (Experimental): Standard of care (SOC)+low dose COVID-HIG. COVID-HIG will be administered via intravenous infusion. once a day, for three consecutive days (Day 0, day 1, and Day 2). And it could be administered again for 1-2 days according to the clinical improvement of subjects, and the total number of infusions should not exceed5 times.
  Interventions: Biological: Human COVID-19 immunoglobulin (pH4) for intravenous injection
- Control Group (Placebo Comparator): Standard of care (SOC)+placebo (0.9% sodium chloride). Placebo will be administered via intravenous infusion. once a day, for three consecutive days (Day 0, day 1, and Day 2). And it could be administered again for 1-2 days according to the clinical improvement of subjects, and the total number of infusions should not exceed5 times.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Human COVID-19 immunoglobulin (pH4) for intravenous injection — The initial infusion rate is 0.01 ~ 0.02 ml/kg body weight/minute (1ml is about 20 drops). If there was no adverse reaction after 15 minutes, the infusion rate could be gradually accelerated. However, it should not exceed 0.08 ml/kg body weight/minute.
  Other Names: COVID-HIG
  Arms: High Dose Group; Low Dose Group
Drug: Placebo — The initial infusion rate is 0.01 ~ 0.02 ml/kg body weight/minute (1ml is about 20 drops). If there was no adverse reaction after 15 minutes, the infusion rate could be gradually accelerated. However, it should not exceed 0.08 ml/kg body weight/minute
  Other Names: 0.9% sodium chloride injection
  Arms: Control Group

SUMMARY:
A randomized, double-blind, placebo-controlled phase II exploratory clinical trial to evaluate the efficacy and safety of Human COVID-19 immunoglobulin (pH4) for intravenous injection (COVID-HIG) in the treatment of patients with COVID-19.

DETAILED DESCRIPTION:
Eligible adault patients with confirmed COVID-19 will be randomized 1:1:1 to receive intravenous injections of High-dose COVID-HIG, Low-dose COVID-HIG or Placebo ( 0.9% sodium chloride injection). Patients in each arm will receive continued standard of care (SOC) therapy. The primary efficacy end point is the median time to clinical improvement (defined as clinical improvement of at least 2 points from baseline on the 7-point ordinal scale) observed from 0 to 28 days after the first administration.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 and <65 years of age when signing the ICF, male or femal.
2. Positive testing by virologic test (SARS-CoV-2 virus nucleic acid test,result of RT-PCR within 3 days are accpetable) before randomization.
3. COVID-19 related clinical symptoms (fever or respiratory symptoms, etc.) progresses before randomization.
4. Inpatients with moderate or severe COVID-19 (severity is graded by FDA standard).
5. With early warning signs for severe/critical cases, meet any of the following indicators: ①Progressive exacerbation of hypoxemia or respiratory distress; ②Deterioration of tissue oxygenation or progressive hyperlactatemia. ③ Rapid decrease in lymphocyte count or steady increase in inflammatory markers such as IL-6, CRP, and ferritin. ④Significant increase of D-dimer and other related indexes of coagulation function. ⑤Chest imaging showing rapid progression of lung lesions.
6. Randomization should be within 10 days of COVID-19 symptoms onset.
7. Subjects (including their partners) have no pregnancy plan and voluntarily take effective contraceptive measures from signing ICF to 3 months after he/she finished the trial.
8. Willing to comply with the requirements, and cooperate when collecting of nasopharyngeal swabs and venous blood for testing according to the protocol; and willing to complete the study.
9. Able to consent, and willing to sign the ICF.

Exclusion Criteria:

1. Asymptomatic infection, mild or critical COVID-19.
2. SP02 < 93% under high-flow oxygen inhalation, or receiving of invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO).
3. Reinfected subjects with historical confirmed COVID-19, detectable by SARS-CoV-2 serological test (nasopharyngeal SARS-CoV-2 RNA levels or serum antibody).
4. May be transferred to another hospital, that is not one of the trial sites, within 72 hours.
5. Meets one of the following high-risk factors: a) Pre-existing cardiovascular (including uncontrolled hypertension: SBP≥ 160 mmHg and/or DBP≥ 100 mmHg) and cerebrovascular diseases, chronic lung diseases (chronic obstructive pulmonary disease (COPD), moderate to severe asthma), diabetes (HbA1c > 9.0%), chronic liver diseases, chronic kidney diseases, malignancies or other complicated diseases. b) Pre-existing Immunosuppression (such as AIDS, long-term use of corticosteroids or other immunosuppressive drugs that lead to a weakened immune function). c) Obesity: body mass index ≥ 35. d) Heavy smokers: ≥20 cigarettes per day on average.
6. History of allergic to IVIG, other plasma proteins or blood products, history of selective IgA deficiency with presence of anti-IgA antibodies.
7. Vaccinated in last 8 weeks, such as influenza, poliomyelitis, measles, rubella, mumps and varicella virus vaccines.
8. May worsen and progress to critical COVID-19 rapidly.
9. Useage of other antiviral drugs to treat SARS-CoV-2 (except the basic treatment specified in the protocol) before randomization.
10. History of major surgery (defined as life-threatening surgery, requiring general anesthesia and causing severe bleeding, including bone and joint surgery on elbow, shoulder, hip, knee, ankle and spine) within 8 weeks before screening (including 8 weeks), or plan to surgery during the trial, which may bring unacceptable risks to the subjects, evaluation by investigators.
11. ALT or AST > 2 times of the normal range upper limit, or Ccr < 60 ml/min.
12. D-dimer increased significantly (> 1 mg/L); History of thromboembolism or coagulation diseases in last 1 year, such as acute coronary syndrome, cerebrovascular syndrome, pulmonary or deep vein thrombosis, etc.
13. Positive of virues makers ( positive of HBsAg, HCV-Ab, or Treponema pallidum specific antibody).
14. History of organ transplantation (such as heart, lung, liver, kidney, etc.
15. Pregnant or lactating female.
16. Other subjects who are not suitable to participate in the trial considered by the investigator, such as potential compliance problems, can not complete all the examinations and evaluations according to the protocol, mental illness, obvious mental disorders; Incapacity or cognitive ability caused by other reasons.
17. History of participated in other investigate drugs or medical devices clinical trials in last 1 month before signing ICF.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2021-12-30 (Estimated); Primary Completion 2023-06-20 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Time to clinical improvement | within 28 days
  The primary efficacy end point is the median time to clinical improvement (defined as clinical improvement of at least 2 points from baseline on the 7-point ordinal scale) observed from 0 to 28 days after the first administration.
  1. Death
  2. Hospitalized, receiving Invasive mechanical ventilation or ECMO
  3. Hospitalized, receiving non-invasive ventilation or high-flow oxygen devices
  4. Hospitalized, requiring Low flow supplemental oxygen
  5. Hospitalized, not requiring oxygen- but receiving ongoing medical care (related or not related to COVID-19)
  6. Hospitalized/not hospitalized, Requiring neither oxygen nor ongoing medical care (other than that specified in the the protocol for COVID-HIG adminstration)
  7. Not hospitalized, discharge or prepare for discharge from a healthcare facility

SECONDARY OUTCOMES:
Changes of 7-point ordinal scale for COVID-19 clinical improvement | 7 days, 14 days, and 28 days
  Compare the clinical status of subjects in each group on day 7, 14, and 28 after the first administration using the primary 7-point ordinal outcome scale. Outcome is reported as the percent of subjects in each of 7 categories and changes in each group compared with baseline.
COVID-19-Related Symptoms | 1 day, 3 days, 5 days, 7 days and 14 days
  Outcome is reported as changes in each group compared with baseline.
Discharge Status | 7 days, 14 days, and 28 days
  Outcome is reported as the percent of subjects in each arm who discharged at day 7, 14, and 28 post treatment.
Length of hospital stay | within 28 days
  Number of days between the first administration and discharge.
All-cause Mortality | within 28 days
  Outcome is reported as the all-cause mortality within 28 days of each arm.
Negativization rate of SARS-CoV-2 nucleic acid | within 72 hrs (24 hrs, 48 hrs, 72 hrs), 7 days, 14 days, and 28 days
  Outcome is reported as the percent of subjects with negative results in each arm.
Changes of leukocyte count, lymphocyte count, C-reactive protein, IL-6 and SARS-CoV-2 nucleic acid (quantitative) | 1 day, 3 days, 5days, 7 days, 14 days
  Outcome is reported as the changes of leukocyte count, lymphocyte count, C-reactive protein, IL-6, and SARS-CoV-2 nucleic acid (quantitative) on 1day, 3days, 5days, 7 days, and 14 days commpared with baseline.
Treatment in ICU | within 28 days
  The proportion and number of subjects who need treatment in ICU within 28 days after the first administration.
SARS-CoV-2 Neutralizing Antibody Level | 1 day, 3 days, 7 days, and 28 days
  Outcome reported as the changes in anti-SARS-CoV-2 neutralizing antibody titer in blood from baseline to 1 day, 3 days, 7 days, and 28 days post treatment. Outcome is reported in units of antibody titer.
Glucocorticoid therapy | within 28 days
  The proportion and the number of subjects receiving glucocorticoid therapy within 28 days after the first administration.
Rate of worsening | within 28 days
  Worsening is defined as the 2 least favorable categories on the primary ordinal scale.
  Outcome is reported as the percent of subjects in each arm who are characterized as worsening within 28 days post treatment.
Finger oxygen saturation | 1 day, 3 days, 5 days, 7 days, 14 days, and 28 days
  Change of finger oxygen saturation compared with the baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Nawal Al Kaabi, MBBA, Principal Investigator — Sheikh Khalifa Medical City, SEHA
Locations (1):
- Al Rahba Hospital, Abu Dhabi, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No